CLINICAL TRIAL: NCT07221006
Title: Investigating the Impact of Facility Dog Intervention on Pediatric Patient Fear, Coping, and Anxiety During Inpatient Admission
Brief Title: Impact of Facility Dog Intervention on Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Sarah Scott, Principal Investigator, Children's Hospital Colorado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-1381
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Inpatients; Pediatric
Keywords: Emotional Support Dog; Pet Therapy Dog; Child Life Specialist; anxiety; fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child life specialist intervention + facility dog led mindfulness (Experimental): Participants will receive a 20-minute mindfulness coping intervention from a CCLS handler and their facility dog. The CCLS will introduce themselves and their facility dog and explain the activity, then implement a guided mindfulness activity while the child holds their hand on the facility dog's stomach/chest.
  Interventions: Behavioral: Mindfulness Activity led by CCLS and Facility Dog
- Child life specialist led mindfulness (Active Comparator): Participants will receive a 20-minute mindfulness coping intervention from a CCLS. The CCLS will introduce themselves and their role and explain the activity and then implement a guided mindfulness activity while the child holds a stress ball.
  Interventions: Behavioral: Mindfulness Activity led by CCLS
- Child life activity coordinator led coloring activity (Other): Participants will complete a 20-minute coloring activity facilitated by a Child Life Activity Coordinator (CLAC). Children aged 8-12 years old will be provided a medical dog coloring sheet with crayons; children aged 13-17 years old will be provided an adult coloring sheet that uses a dog image and colored pencils.
  Interventions: Behavioral: Coloring page activity led by CLAC

INTERVENTIONS:
Behavioral: Coloring page activity led by CLAC — Participants will be provided coloring pages and colored pencils or crayons led by a Child Life Activity Coordinator, and will engage in the activity for 15 minutes.
  Arms: Child life activity coordinator led coloring activity
Behavioral: Mindfulness Activity led by CCLS — Participants will engage in a 10 minute mindfulness activity led by a Certified Child Life Specialist who will follow a mindfulness script. Participants will hold a stress ball during the activity.
  Arms: Child life specialist led mindfulness
Behavioral: Mindfulness Activity led by CCLS and Facility Dog — Participants will engage in a 10 minute mindfulness activity led by a Certified Child Life Specialist who will follow a mindfulness script. Participants will be able to be next to and touch the medical dog during the activity.
  Arms: Child life specialist intervention + facility dog led mindfulness

SUMMARY:
The goal of this clinical trial is to learn if medical dog intervention facilitated by a Certified Child Life Specialist (CCLS) impacts pediatric patient coping, fear, and anxiety during inpatient admissions. The main questions it aims to answer are:

What impact does facility dog support via a CCLS have on patient fear, coping, and anxiety? What effect does facility dog support via a CCLS have on patient heart rate? Researchers will compare medical dog intervention facilitated by a CCLS, CCLS intervention, and a coloring activity to see if medical dog interventions positively impact coping, fear, and anxiety.

Participants will:

Receive a visit from a medical dog and their CCLS handler, a CCLS, or a Child Life Activity coordinator.

Engage in a mindfulness or coloring activity. Answer surveys regarding anxiety, coping, and fear. Have their heart rate measured before, during, and after their assigned intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to an inpatient unit at Children's Hospital Colorado Anschutz Medical Campus
* Who are eight to 17 years old.

Exclusion Criteria:

* Isolation precautions
* Primary reason for admission is due to suicidality, self-injurious behavior, or injurious behavior
* Patients with history of or currently presenting with aggression or unsafe behavior
* Severe comorbidities secondary to traumatic brain injury, neurological disorder or neurodevelopmental issues that may confound study outcomes and administration of the study protocol (e.g., intellectual disability)
* Not medically stable
* Have a fear of dogs
* Have an allergy to dogs
* Have had a visit from a medical dog and medical dog handler during their current admission
* Patient has an urgent or time-sensitive need requiring medical dog support - Patient is non-verbal.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Spielberger State Trait Anxiety Inventory Short Form | Baseline and approximately 15 minutes after starting the intervention.
  A 6-item measure that assesses anxiety via self-report. Individuals rate their agreement with six statements on a 4-point scale, ranging from 1 (not at all) to 4 (very much), with higher scores indicating more anxiety.
Children's Fear Scale | Baseline and approximately 15 minutes after starting the intervention.
  A 1-item measure that assesses fear via self-report faces scale. Individuals rate their fear on a scale, ranging from no fear to extreme fear, by selecting one of five face pictures that matches how they feel.
Coping Questionnaire - Child | Approximately 15 minutes after starting the intervention.
  Measures youth's perceived ability to cope on a three-item, individualized measure. Children rate their ability to make themselves less upset during an anxiety-provoking situation on a 7-point scale, ranging from 1 (not at all able to help myself or him/herself) to 7, with lower scores indicating poor coping.

SECONDARY OUTCOMES:
Heart Rate | Baseline, before the intervention, 5 minutes after intervention start, post-intervention (approximately 15 minutes after intervention start).
  Participants' heart rate will be measured at four time points using a bedside heart rate monitor.
Parent Survey | Before the intervention.
  Legal guardians will be if the participant has any developmental and/or psychological diagnoses, as well as if the patient has a dog at home.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Scott, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided